CLINICAL TRIAL: NCT04732403
Title: The Effect of Patient Positioning on Ureteral Efflux During Intraoperative Cystoscopy: a Randomized Controlled Trial
Brief Title: Ureteral Jets and Patient Positioning Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arizona (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2011188102
Record Dates: First submitted 2021-01-27; First posted 2021-02-01 (Actual); Last update posted 2024-11-01 (Actual); Status verified 2021-06

CONDITIONS: Ureteral Injury; Surgery--Complications
Keywords: ureteral injury; cystoscopy; hysterectomy; gynecologic surgery
MeSH Terms: interventions — Patient Positioning

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 0 degree supine position (No Intervention): Surgical bed will be set to a 0 degree supine position
- 10-20 degree angle in reverse Trendelenburg (Experimental): Surgical bed will be set to a 10-20 degree angle in reverse Trendelenburg
  Interventions: Other: Patient Position

INTERVENTIONS:
Other: Patient Position — The patient will be placed in an angle on the surgical table during cystoscopy.
  Arms: 10-20 degree angle in reverse Trendelenburg

SUMMARY:
The objective of the study is to identify the relationship between patient position during surgery and time to confirmation of ureteral patency on cystoscopy.

DETAILED DESCRIPTION:
Patients will be randomized to one of two arms: 0 degree supine position and 10-20 degree angle in reverse Trendelenburg. Our working hypothesis is that positioning a patient in 10-20 degree angle reverse Trendelenburg will result in shorter time to confirmation of bilateral ureteral patency and shorter total cystoscopy time, without a change in delayed diagnosis of ureteric injury.

Primary outcome: time to confirmation of bilateral ureteral patency Secondary outcome: total cystoscopy time, need for alternative modalities to aid in ureteral efflux visualization, delayed diagnosis of ureteric injury (evaluated 6 weeks postoperatively via chart review)

ELIGIBILITY:
Inclusion Criteria:

1. Female patients
2. Greater than or equal to 18 years old
3. English-speaking
4. Scheduled benign gynecologic or urogynecologic surgery in which routine cystoscopy at Banner University Medical Center - Phoenix; Dr. Mourad, Dr. Mahnert or Dr. Rachael Smith.

Exclusion Criteria:

1. Patients with underlying chronic kidney disease (creatinine <1)
2. Known renal anomaly such as prior surgical removal of a kidney or underlying ureteral obstruction
3. Current ureteral stent in place,
4. Pregnancy,
5. Contraindication to any of the interventions (i.e., documented allergies)

Ages: 18 Years to 89 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
time to confirmation of bilateral ureteral patency | 1 day
  time between initiation of cystoscopy and visualization of second ureteral jet in minutes

SECONDARY OUTCOMES:
total cystoscopy time | 1 day
  Total time of cystoscopy
need for alternative modalities to aid in ureteral efflux visualization | 1 day
  After 10 minutes of no jet, it is okay for the surgeon to use alternative methods, including dextrose, sodium fluorescein, indigo carmine, IV diuretics, etc.
delayed diagnosis of ureteric injury | 6 weeks after surgery
  evaluated 6 weeks postoperatively via chart review

CONTACTS AND LOCATIONS:
Overall Officials: Jamal Mourad, DO, Principal Investigator — University of Arizona
Locations (1):
- Banner University Medical Center Phoenix, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Teeluckdharry B, Gilmour D, Flowerdew G. Urinary Tract Injury at Benign Gynecologic Surgery and the Role of Cystoscopy: A Systematic Review and Meta-analysis. Obstet Gynecol. 2015 Dec;126(6):1161-1169. doi: 10.1097/AOG.0000000000001096. PMID 26551173
- [Background] Vakili B, Chesson RR, Kyle BL, Shobeiri SA, Echols KT, Gist R, Zheng YT, Nolan TE. The incidence of urinary tract injury during hysterectomy: a prospective analysis based on universal cystoscopy. Am J Obstet Gynecol. 2005 May;192(5):1599-604. doi: 10.1016/j.ajog.2004.11.016. PMID 15902164
- [Background] Gilmour DT, Baskett TF. Disability and litigation from urinary tract injuries at benign gynecologic surgery in Canada. Obstet Gynecol. 2005 Jan;105(1):109-14. doi: 10.1097/01.AOG.0000144127.78481.8c. PMID 15625150
- [Background] Delacroix SE Jr, Winters JC. Urinary tract injuries: recognition and management. Clin Colon Rectal Surg. 2010 Sep;23(3):221. doi: 10.1055/s-0030-1263063. No abstract available. PMID 21886472
- [Background] Brandes S, Coburn M, Armenakas N, McAninch J. Diagnosis and management of ureteric injury: an evidence-based analysis. BJU Int. 2004 Aug;94(3):277-89. doi: 10.1111/j.1464-410X.2004.04978.x. No abstract available. PMID 15291852
- [Background] Cohen SA, Carberry CL, Smilen SW. American Urogynecologic Society Consensus Statement: Cystoscopy at the Time of Prolapse Repair. Female Pelvic Med Reconstr Surg. 2018 Jul/Aug;24(4):258-259. doi: 10.1097/SPV.0000000000000529. PMID 29369837
- [Background] Kim JH. Urogynecology and Reconstructive Pelvic Surgery. 4th ed. Int Neurourol J. 2015 Mar;19(1):51. doi: 10.5213/inj.2015.19.1.51. No abstract available. PMID 25833482
- [Background] AAGL Advancing Minimally Invasive Gynecology Worldwide. AAGL Practice Report: Practice guidelines for intraoperative cystoscopy in laparoscopic hysterectomy. J Minim Invasive Gynecol. 2012 Jul-Aug;19(4):407-11. doi: 10.1016/j.jmig.2012.05.001. PMID 22748947
- [Derived] Galhotra S, Zeng K, Hu C, Norton T, Mahnert N, Smith R, Mourad J. The Effect of Patient Positioning on Ureteral Efflux During Intraoperative Cystoscopy: A Randomized Controlled Trial. J Minim Invasive Gynecol. 2023 Jan;30(1):13-18. doi: 10.1016/j.jmig.2022.09.003. Epub 2022 Sep 11. PMID 36103970